CLINICAL TRIAL: NCT03207152
Title: Biomarkers Predicting Infectivity in an Experimental Human Influenza Model
Acronym: PRESAGE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Imperial College of London (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00082500
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Influenza A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Influenza A/California/04/2009 (Experimental): Participants will be inoculated with Influenza A/California/04/09 3.5x10(4) tissue culture infective dose 50% (TCID50) in 1 mL in Dulbecco's phosphate buffered saline (DPBS) delivered by intranasal drops. They will then be monitored as in-patients for 10 days with daily clinical assessment and blood and respiratory tract sampling. Following discharge, they will be followed up for up to 6 months post-inoculation.
  Interventions: Biological: Influenza A/California/04/09

INTERVENTIONS:
Biological: Influenza A/California/04/09 — Good Manufacturing Practices-certified Influenza A/California/04/09 3.5x10(4) TCID50 in 1 mL in DPBS delivered by intranasal drops

SUMMARY:
This study aims to test the hypothesis that gene transcriptional changes occur within 24 hours of virus exposure in the blood and nasal mucosa, and to identify early biomarker signatures that are predictive of higher viral shedding at the peak of disease

DETAILED DESCRIPTION:
This study will systematically investigate the early pre-symptomatic period following exposure to influenza in humans. The data obtained will be essential for further understanding of the natural history of human antiviral responses, and will allow us to identify a panel of biomarkers that can predict which individuals will go on to more severe symptoms and higher viral shedding, so that treatments and other interventions can be made at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 18 to 55 years, able to give informed consent

Exclusion Criteria:

* Chronic respiratory disease (asthma, chronic obstructive pulmonary disease, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 6 months
* Acute upper respiratory infection or sinusitis in the past 6 weeks
* Smoking in the past 6 months OR >5 pack-year lifetime history
* Subjects with allergic symptoms present at baseline
* Clinically relevant abnormality on chest X-ray
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Subjects with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* Known immunoglobulin A deficiency, immotile cilia syndrome, or Kartagener's syndrome
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by the study doctor to make the participant unsuitable for the study
* Pregnant or breastfeeding women
* Positive urine drug screen
* Detectable baseline haemagglutination inhibition titres against influenza challenge strains
* History of hypersensitivity to eggs, egg proteins, gentamicin, gelatin or arginine, or with life-threatening reactions to previous influenza vaccinations

All women of childbearing age will have a pregnancy test performed prior to virus inoculation to exclude pregnancy and be required to use contraception throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Viral load | 28 days
  Nasal wash viral load by quantitative polymerase chain reaction (qPCR)

SECONDARY OUTCOMES:
Symptoms | 28 days
  Self-reported upper and lower respiratory and systemic symptoms by diary card
Differentially expressed genes in blood | 9 months
  Differentially expressed genes analysed by RNA sequencing of whole blood
Differentially expressed genes in nasal curettage | 9 months
  Differentially expressed genes analysed by RNA sequencing of nasal curettage samples
Metabolomics in serum | 9 months
  Differentially expressed metabolites in serum by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, BMBCh PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Duke university, such as ethnicity and age. It will be identifiable only by their unique study code, with no personal details.